CLINICAL TRIAL: NCT02882204
Title: Tracking Outcomes in Psychosis
Acronym: TOPSY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 10014067
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- First Episode Patients: First episode patients new to the PEPP program.
- Chronic Patients: Existing patients who have been enrolled in the PEPP program for >3 years
- Healthy Controls: Healthy controls who are not currently in treatment for any major mental illness defined using DSM-V criteria.
- Cliniucal High Risk patients: Patients who are accessing PEPP services during the prodromal phase of psychotic illness.

SUMMARY:
The investigators propose to study the brain processes that result in thought and language disorder and influence outcomes seen in patients with schizophrenia using a combination of brain scans and clinical assessments. The project will assess patients at various stages of psychosis (Clinical high risk, first episode and chronic stage >3 years of illness) referred to the Prevention and Early Intervention in Psychosis Programme using Magnetic Resonance Imaging (MRI scans). To track the outcome of this illness, investigators will follow-up patients over 3 years and collect MRI scans over four sessions for each first episode patient, and two sessions for clinical high risk patients, chronic patients, and healthy controls. Participants will also complete a clinical assessment examining symptoms and functioning as per the current clinical practice within the PEPP program at each scanning session.

DETAILED DESCRIPTION:
OBJECTIVES: The objective of this study is to investigate the pathophysiology of Formal Thought Disorder and variable outcomes in the early stages of schizophrenia. In particular, investigators aim to test the hypothesis that 1. Anatomical abnormalities involving the grey matter of the Anterior Insula and Medial Prefrontal Cortex in first episode schizophrenia predicts FTD that persists by 6 months of illness 2. An excess of glutamine/glutamate, or reduction in glutathione, in Medial Prefrontal Cortex at index episode will be associated with persistent FTD 3.Aberrant connectivity between Anterior Insula and Medial Prefrontal Cortex will specifically predict the severity of persistent FTD irrespective of the stage of illness; the change in this connectivity will track the variable 3-year outcome among patients with first episode of psychosis.

METHODS: This study will employ a cross-sectional design recruiting n=126 participants from the Prevention & Early Intervention Program for Psychoses (PEPP). Four groups of participants will be assessed: patients at a later stage of schizophrenia (chronic illness group) (n=42), newly referred first episode group of PEPP patients (n=84), Clinical High Risk patients (n=60) and healthy Controls (n=45). Measurements: Patients will be diagnosed using the criteria for schizophrenia according to DSM-V(34). Demographic variables such as age, gender and parental socioeconomic status will be recorded to adjust for potential confounding effects. Patients will undergo baseline assessments to assess seven features of FTD (poverty of speech, weakening of goal, perseveration, looseness, peculiar word usage, peculiar sentence usage and peculiar logic) in line with the validated procedure for administering Thought Language Index [TLI](17). First episode patients will undergo four 7T MRI scanning sessions over the course of 2.5 years (baseline, 6 months, 18 months, 30 months)lasting for 60 minutes each, as described in our previous work (15). During this time, researchers will perform MR spectroscopy (MPFC voxel (31)), T1 weighted structural scan and eyes-closed, task-free, 6 minutes resting-state functional MRI. 6 months after the onset of first episode, the clinical assessment will be repeated using TLI. Patients with persistent FTD will be identified (from previous studies, 40% of patients are expected to have persistent FTD (9)) and separated from patients who have no FTD at 6-months time point. Patients with established illness will undergo only 2 scans: baseline and 1 year later.

ELIGIBILITY:
Inclusion Criteria:

* 16-45 years old
* Outpatient of the Prevention and Early Intervention Program for Psychosis

Exclusion Criteria:

* Drug or alcohol dependence in past year
* History of head injury (with associated unconsciousness for any period)
* Mental retardation or suffering from medical conditions such as untreated hypertension, diabetes, hepatic/renal insufficiency, neurological illnesses
* Otherwise unable to provide informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population includes two groups of individuals:
  1. First Episode psychotic patients: This group will contain 84 new patients enrolled in the Prevention and early Intervention Program for Psychosis.
  2. Chronic Patients: This group will contain 42 patients who have been enrolled in the Prevention and Early Intervention Program for Psychosis for >3 years.
  3. Healthy Controls: This group will contain 42 healthy controls not being treated for a major mental illness defined using DSM-V criteria.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Thought Language Index Score between baseline and 6 months | 6 Months
  Predicting the change in TLI score based on baseline anatomical abnormalities identified through MRI
Time to remission of positive symptoms of psychosis | 30 months
  The time between baseline and remission of positive symptoms based on PANSS-8
Time to remission of negative symptoms of psychosis | 30 months
  The amount of time between baseline and remission of negative symptoms based on PANSS-8
Emergence of treatment resistance using operational criteria | 30 months

SECONDARY OUTCOMES:
Change in Thought Language Index score between baseline and longitudinal follow up-dates (12 months, 18 months, 24 months and 30 months) | 1-2.5 years
  Net change in TLI score as predicted by anatomical abnormalities associated with imaging at various imaging time points.
Change in overall symptoms over time | 30 months
  Tracking changes in scores on the PANSS-8 over the 30 months of follow up for first episode patients
Changes in myelin content | 30 months (follow up period for first episode patients)
  Longitudinal changes in myelin content as measured using quantitative t1 images

CONTACTS AND LOCATIONS:
Locations (1):
- Robarts Research, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrow M, Marengo JT. Schizophrenic thought disorder at followup: its persistence and prognostic significance. Schizophr Bull. 1986;12(3):373-93. doi: 10.1093/schbul/12.3.373. PMID 3764358
- [Background] Palaniyappan L, Mahmood J, Balain V, Mougin O, Gowland PA, Liddle PF. Structural correlates of formal thought disorder in schizophrenia: An ultra-high field multivariate morphometry study. Schizophr Res. 2015 Oct;168(1-2):305-12. doi: 10.1016/j.schres.2015.07.022. Epub 2015 Jul 29. PMID 26232240
- [Background] Liddle PF, Ngan ET, Caissie SL, Anderson CM, Bates AT, Quested DJ, White R, Weg R. Thought and Language Index: an instrument for assessing thought and language in schizophrenia. Br J Psychiatry. 2002 Oct;181:326-30. doi: 10.1192/bjp.181.4.326. PMID 12356660
- [Background] Aoyama N, Theberge J, Drost DJ, Manchanda R, Northcott S, Neufeld RW, Menon RS, Rajakumar N, Pavlosky WF, Densmore M, Schaefer B, Williamson PC. Grey matter and social functioning correlates of glutamatergic metabolite loss in schizophrenia. Br J Psychiatry. 2011 Jun;198(6):448-56. doi: 10.1192/bjp.bp.110.079608. PMID 21628707
- [Background] American Psychiatric Association, Diagnostic and Statistical Manual of Mental Disorders (DSM-5®) (2013).